CLINICAL TRIAL: NCT04915807
Title: A Prospective Study for Real-world Data (RWD) of Ramucirumab Plus Paclitaxel in Patients With Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Real-world Data (RWD) of Ramucirumab Plus Paclitaxel
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Zang, Dae Young, Professor, Hallym University Medical Center
Other Study IDs: KCSG ST21-06
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: Real-world data; Gastric cancer; Gastroesophageal junction adenocarcinoma; Ramucirumab; Paclitaxel; Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ramucirumab; Paclitaxel; taxane; Irinotecan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective population: The target group for the purpose of prospectively collecting the clinical data (RWD) of patients using ramucirumab/paclitaxel as 2nd-line chemotherapy in patients with locally advanced unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma
  Interventions: Drug: Ramucirumab and paclitaxel
- Historical retrospective population: The target group for the purpose of retrospectively collecting the clinical data (RWD) of patients who have failed platinum-based palliative first-line therapy, and who started the following second-line therapy: taxane, irinotecan , or fluoropyrimidine-based single or combined chemotherapy, before May 1, 2018, when health insurance coverage for the ramucirumab/paclitaxel combination therapy started in South Korea.
  Interventions: Drug: Taxane, irinotecan, or fluoropyrimidine-based single or combined chemotherapy

INTERVENTIONS:
Drug: Ramucirumab and paclitaxel — Ramucirumab/paclitaxel as a second-line chemotherapy after May 1, 2018, when health insurance coverage for the combination therapy started
  Other Names: Prospective population
  Groups: Prospective population
Drug: Taxane, irinotecan, or fluoropyrimidine-based single or combined chemotherapy — Taxane, irinotecan , or fluoropyrimidine-based single or combined chemotherapy as a second-line therapy
  Other Names: Historical retrospective population
  Groups: Historical retrospective population

SUMMARY:
Real World Data (RWD) obtained from real clinical sites is data obtained after administering a drug to patients with different characteristics in daily practice, and Real World Evidence (RWE) is established based on RWD. It is possible to overcome the disadvantage of RCT, which cannot reflect all the various variables in the actual clinical field as it is conducted for only subset of patients.

Researchers planned to prospectively collect RWD of ramucirumab/paclitaxel combination therapy as 2nd-line chemotherapy in patients with locally advanced unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
Most drugs are introduced into the medical market based on efficacy derived from randomized controlled trials (RCTs) in a subset of patient groups in which the age, presence of comorbidities, and general conditions of the target patient are strictly controlled by the researcher.

Real World Data (RWD) obtained from real clinical sites is data obtained after administering a drug to patients with different characteristics in daily practice, and Real World Evidence (RWE) is established based on RWD. It is possible to overcome the disadvantage of RCT, which cannot reflect all the various variables in the actual clinical field as it is conducted for only subset of patients.

Researchers have collected retrospective RWD from patients who used ramucirumab/paclitaxel in a previous study (KCSG ST19-16). Considering the limitations of RWD obtained through retrospective data collection, it is necessary to generate RWE through RWD, which prospectively collects various clinical data obtained in the process of using new anticancer drugs.

ELIGIBILITY:
1. Prospective population

   Inclusion Criteria:
   * Patients aged 19 years or older and histologically or cytologically confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma
   * Patients with locally advanced or metastatic disease for which curative resection is not possible.
   * Patients who have failed fluoropyrimidine and platinum (cisplatin or oxaliplatin)-based chemotherapy as palliative first-line therapy
   * Patients who is starting ramucirumab/paclitaxel combination therapy after the study initiation date

   Exclusion Criteria:
   * Patients receiving ramucirumab monotherapy
   * Patients receiving ramucirumab/paclitaxel in clinical trial or receiving without being covered by health insurance
   * Patients unable to communicate or incapable of understanding documents for patient report outcomes
2. Historical retrospective population

Inclusion Criteria:

* Patients aged 19 years or older and histologically or cytologically confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma
* Patients with locally advanced or metastatic disease for which curative resection is not possible
* Patients who have failed platinum-based palliative first-line therapy, and who started the following second-line therapy: taxane, irinotecan , or fluoropyrimidine-based single or combined chemotherapy, before May 1, 2018

Exclusion Criteria:

* Patients receiving ramucirumab monotherapy
* Patients receiving ramucirumab/paclitaxel in clinical trial or receiving without being covered by health insurance

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting university hospitals located in major cities in South Korea
Sampling Method: Non-Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Until September 30, 2023
  Time from the start of ramucirumab/paclitaxel to death from any cause
Progression-free survival | Until September 30, 2023
  Time from the start of ramucirumab/paclitaxel to disease progression or death from any cause

SECONDARY OUTCOMES:
Incidence of adverse events | Until September 30, 2023
  Number (percentage) of subjects reporting adverse events according to CTCAE v5.0
Time to progression | Until September 30, 2023
  Time from the start of ramucirumab/paclitaxel to disease progression
Objective response rate | Until September 30, 2023
  The proportion of subjects confirmed complete or partial response according to RECIST v1.1
Disease control rate | Until September 30, 2023
  The proportion of subjects confirmed complete response, partial response or stable disease according to RECIST v1.1
Duration of response | Until September 30, 2023
  Time from documentation of tumor response to disease progression
Adverse events of special interest | Until September 30, 2023
  Number (percentage) of subjects reporting adverse events of special interest associated with ramucirumab/paclitaxel: hypertension, proteinuria, gastrointestinal bleeding or perforation, delayed wound healing, deep vein thrombosis, arterial thrombosis, stroke according to on CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, Principal Investigator — Hallym University Medical Center
Locations (9):
- South Korea (9):
  - Hallym University Sacred Heart Hospital, Anyang
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Seoul National University Bundang Hospital, Seongnam
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jung KW, Won YJ, Kong HJ, Lee ES. Cancer Statistics in Korea: Incidence, Mortality, Survival, and Prevalence in 2016. Cancer Res Treat. 2019 Apr;51(2):417-430. doi: 10.4143/crt.2019.138. Epub 2019 Mar 18. PMID 30913865
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Wagner AD, Grothe W, Haerting J, Kleber G, Grothey A, Fleig WE. Chemotherapy in advanced gastric cancer: a systematic review and meta-analysis based on aggregate data. J Clin Oncol. 2006 Jun 20;24(18):2903-9. doi: 10.1200/JCO.2005.05.0245. PMID 16782930
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Kim HS, Kim HJ, Kim SY, Kim TY, Lee KW, Baek SK, Kim TY, Ryu MH, Nam BH, Zang DY. Second-line chemotherapy versus supportive cancer treatment in advanced gastric cancer: a meta-analysis. Ann Oncol. 2013 Nov;24(11):2850-4. doi: 10.1093/annonc/mdt351. Epub 2013 Aug 13. PMID 23942775
- [Background] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Background] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Background] Smyth EC, Verheij M, Allum W, Cunningham D, Cervantes A, Arnold D; ESMO Guidelines Committee. Gastric cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2016 Sep;27(suppl 5):v38-v49. doi: 10.1093/annonc/mdw350. No abstract available. PMID 27664260
- [Background] Muro K, Van Cutsem E, Narita Y, Pentheroudakis G, Baba E, Li J, Ryu MH, Zamaniah WIW, Yong WP, Yeh KH, Kato K, Lu Z, Cho BC, Nor IM, Ng M, Chen LT, Nakajima TE, Shitara K, Kawakami H, Tsushima T, Yoshino T, Lordick F, Martinelli E, Smyth EC, Arnold D, Minami H, Tabernero J, Douillard JY. Pan-Asian adapted ESMO Clinical Practice Guidelines for the management of patients with metastatic gastric cancer: a JSMO-ESMO initiative endorsed by CSCO, KSMO, MOS, SSO and TOS. Ann Oncol. 2019 Jan 1;30(1):19-33. doi: 10.1093/annonc/mdy502. PMID 30475956
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2014 (ver. 4). Gastric Cancer. 2017 Jan;20(1):1-19. doi: 10.1007/s10120-016-0622-4. Epub 2016 Jun 24. No abstract available. PMID 27342689
- [Background] Guideline Committee of the Korean Gastric Cancer Association (KGCA), Development Working Group & Review Panel. Korean Practice Guideline for Gastric Cancer 2018: an Evidence-based, Multi-disciplinary Approach. J Gastric Cancer. 2019 Mar;19(1):1-48. doi: 10.5230/jgc.2019.19.e8. Epub 2019 Mar 19. No abstract available. PMID 30944757
- [Background] Signorovitch JE, Sikirica V, Erder MH, Xie J, Lu M, Hodgkins PS, Betts KA, Wu EQ. Matching-adjusted indirect comparisons: a new tool for timely comparative effectiveness research. Value Health. 2012 Sep-Oct;15(6):940-7. doi: 10.1016/j.jval.2012.05.004. PMID 22999145
- [Background] Signorovitch JE, Wu EQ, Yu AP, Gerrits CM, Kantor E, Bao Y, Gupta SR, Mulani PM. Comparative effectiveness without head-to-head trials: a method for matching-adjusted indirect comparisons applied to psoriasis treatment with adalimumab or etanercept. Pharmacoeconomics. 2010;28(10):935-45. doi: 10.2165/11538370-000000000-00000. PMID 20831302
- See also: Gastric Cancer: NCCN Guidelines Version 2.2021 — https://www.nccn.org/guidelines/guidelines-detail?category=1&id=1434